CLINICAL TRIAL: NCT00098514
Title: A Phase I Study Of PT523 In Patients With Solid Tumors
Brief Title: Talotrexin in Treating Patients With Advanced or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Geoffrey Shapiro, MD, PhD, Director, Early Drug Development Center, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-183; P30CA006516 (NIH); CDR0000400150; NCI-6400; DFCI-IRB-03183; HANABIO-DFCI-02000
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Intervention Model Description: There were 7 potential PT523 single agent dose levels to be evaluated in this phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Dose Level 1a (Experimental): 10 mg/m2 dose of PT523 administered day 1 of a 28-day cycle as a 5 minute IV infusion (IV bolus)
  Interventions: Drug: talotrexin ammonium
- Dose Level 1b (Experimental): 5 mg/m2 dose of PT523 administered days 1 and 8 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium
- Dose Level 1c (Experimental): 3.33 mg/m2 dose of PT523 administered days 1, 8 and 15 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium
- Dose Level 2 (Experimental): 5 mg/m2 dose of PT523 administered days 1, 8 and 15 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium
- Dose Level 3 (Experimental): 7.5 mg/m2 dose (or 6.7 mg/m2 depending on observed toxicity) of PT523 administered days 1, 8 and 15 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium
- Dose Level 4 (Experimental): 11.25 mg/m2 dose (or 9 mg/m2 depending on observed toxicity) of PT523 administered days 1, 8 and 15 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium
- Dose Level 5 (Experimental): 17 mg/m2 dose (or 12 mg/m2 depending on observed toxicity) of PT523 administered days 1, 8 and 15 of a 28-day cycle as a 5 minute IV infusion
  Interventions: Drug: talotrexin ammonium

INTERVENTIONS:
Drug: talotrexin ammonium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as talotrexin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying side effects, best way to give, and best dose of talotrexin in treating patients with advanced or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of talotrexin in patients in patients with advanced or recurrent solid tumors.
* Determine the safety of this drug in these patients.
* Determine the dose-limiting toxic effects of this drug in these patients.

Secondary

* Determine the pharmacokinetics of this drug in these patients.
* Correlate pharmacokinetic parameters of this drug or patient characteristics with drug-related toxicity in these patients.
* Determine, preliminarily, the antitumor efficacy of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive talotrexin IV over 5 minutes on day 1 OR days 1 and 8 OR days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of talotrexin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 6-10 patients are treated at the MTD.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 9-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignant solid tumor

  * Metastatic or inoperable disease
* No known curative or survival-prolonging palliative therapy exists OR failed these prior therapies
* No leukemia
* No primary CNS tumor
* No third-space fluid collection (i.e., pleural effusion, ascites)

  * Clinically insignificant small pleural or peritoneal effusions identified by CT scan, MRI, or other diagnostic test allowed
* No active* brain metastases, including the following:

  * Evidence of cerebral edema by CT scan or MRI
  * Progression since prior imaging study
  * Requirement for steroids
  * Clinical symptoms of/from brain metastases NOTE: *Treated and/or stable brain metastasis allowed provided patient is asymptomatic

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 2 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* RBC folate ≥ lower limit of normal

Hepatic

* Bilirubin normal
* SGOT and SGPT ≤ 2.5 times upper limit of normal

Renal

* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other uncontrolled serious medical or psychiatric illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior bone marrow transplantation

Chemotherapy

* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior surgery

Other

* Recovered from prior therapy
* More than 3 weeks since prior antifolate therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Paul Eder, MD, Principal Investigator
Locations (1):
- Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts, United States